CLINICAL TRIAL: NCT03330509
Title: Effectiveness of the Supportive and Palliative Care Review Kit (SPARK) for Cancer Patients in the Acute Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Singapore General Hospital (Other); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: NRSMFSP17101
Record Dates: First submitted 2017-10-18; First posted 2017-11-06 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Health Services Research
Keywords: Palliative care; Consultation model

STUDY DESIGN:
Intervention Model Description: A stepped-wedge design will be used for this study, unblinded due to practical challenges of blinding. There will be 4 teams (clusters) within the DMO inpatient service, each comprising a team of senior consultant physicians, middle level and junior doctors, and oncology nurses. This follows current team structures. During the intervention period, a palliative care physician and nurse will join the team as integrated members.
  The study will be conducted over 20 months from November 2017 to June 2019, with each cluster crossing over from 'usual care' to 'spark intervention' at 4-month intervals. Each cluster will be randomly assigned a specific timing of crossing over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cluster 1 (Experimental): Control: 1-4 months; SPARK intervention: 5-20 months
  Interventions: Other: SPARK intervention
- Cluster 2 (Experimental): Control: 1-8 months; SPARK intervention: 9-20 months
  Interventions: Other: SPARK intervention
- Cluster 3 (Experimental): Control: 1-12 months; SPARK intervention: 13-20 months
  Interventions: Other: SPARK intervention
- Cluster 4 (Experimental): Control: 1-16 months; SPARK intervention: 17-20 months
  Interventions: Other: SPARK intervention

INTERVENTIONS:
Other: SPARK intervention — An integrated model of care (SPARK care) in which the palliative care team co-rounds with the medical oncology team, supporting them in their delivery of basic palliative care, seamlessly stepping in and out to deliver specialist palliative care directly to patients when needed.

SUMMARY:
Introduction

There is a rising need for palliative care services in Singapore due to a rapidly ageing population and an increasing incidence of cancer. Current existing resources are inadequate - novel models of care are needed to expand access to palliative care without requiring significantly more specialist palliative care manpower.

Oncologist-driven referrals to a palliative care consultation service is the norm worldwide, including Singapore. This results in variable access to palliative care due to differences in referral practices. Palliative care involvement is also often delayed. In this study, the investigators propose to test Supportive and Palliative care Review Kit (SPARK) - a novel integrated model of care in which the palliative care team co-rounds with the medical oncology team.

Specific Aims and Hypothesis

This study aims to evaluate the impact of SPARK compared to usual care. The study investigators hypothesize that SPARK will result in more advanced cancer patients having access to palliative care, and at the same time operate at lower net cost. The study investigators also hypothesize that the improved efficiency of SPARK will result in shorter hospital length of stay for stage 4 cancer patients.

Methods

A cluster randomized trial with step wedged design will be used to compare SPARK to usual care. Data will be collected on health services utilization and access to palliative care services. Net costs will also be compared between SPARK and usual care. Semi-structured interviews with patients and healthcare professionals will be used to explore differences in experiences of healthcare provision between both models of care.

Importance

Singapore has a rising prevalence of cancer patients who require palliative care input, but only a minority are able to access it at present. If the SPARK model of care proves to be a scalable and cost-effective way of expanding access to palliative care, more cancer patients can benefit from palliative care.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted under the care of the medical oncology team in Singapore General Hospital will be included.

Exclusion Criteria:

* Patients below 21 years old.

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7514 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | 6 months
  Dates of hospital admission and discharge will be collected to measure hospital length of stay

SECONDARY OUTCOMES:
Number of days from hospital discharge to hospital readmission | 30 days
  Date of hospital discharge and date of subsequent hospital admission, if any, will be collected to measure this outcome
Referral to palliative care services | 6 months
  Presence of referral to hospital palliative care consult service, home hospice or other palliative care services will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Centre Singapore, Singapore, Singapore

REFERENCES:
- [Background] Nickolich MS, El-Jawahri A, Temel JS, LeBlanc TW. Discussing the Evidence for Upstream Palliative Care in Improving Outcomes in Advanced Cancer. Am Soc Clin Oncol Educ Book. 2016;35:e534-8. doi: 10.1200/EDBK_159224. PMID 27249764
- [Background] Hui D, Bruera E. Models of integration of oncology and palliative care. Ann Palliat Med. 2015 Jul;4(3):89-98. doi: 10.3978/j.issn.2224-5820.2015.04.01. PMID 26231806
- [Derived] Yang GM, Zhou S, Xu Z, Goh SS, Zhu X, Chong DQ, Tan DS, Kanesvaran R, Yee AC, Neo PS, Cheung YB. Comparing the effect of a consult model versus an integrated palliative care and medical oncology co-rounding model on health care utilization in an acute hospital - an open-label stepped-wedge cluster-randomized trial. Palliat Med. 2021 Sep;35(8):1578-1589. doi: 10.1177/02692163211022957. PMID 34524044

DOCUMENTS (2):
  • Study Protocol (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03330509/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03330509/SAP_001.pdf